CLINICAL TRIAL: NCT00333463
Title: Compliance With Once Daily Glaucoma Medication
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Collaborators: Johns Hopkins University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CMS-06-03
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2010-03

CONDITIONS: Compliance
MeSH Terms: conditions — Patient Compliance | interventions — Methods

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Intervention group: The intervention group watched an educational video, reviewed current barriers to drop-taking and possible solutions with a study coordinator, received regular phone call reminders, and had audible and visible reminders activated on their DA devices.
  Interventions: Behavioral: Intervention
- Non-Intervention Group: The control group was told to take drops as prescribed and received no additional intervention.

INTERVENTIONS:
Behavioral: Intervention — The intervention group watched an educational video, reviewed current barriers to drop-taking and possible solutions with a study coordinator, received regular phone call reminders, and had audible and visible reminders activated on their DA devices.
  Groups: Intervention group

SUMMARY:
A study to examine patient compliance with once daily glaucoma medication

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or ocular hypertension patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary open angle glaucoma or ocular hypertension patients
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Friedman, MD, Study Director — Study Director
Locations (1):
- Ft. Worth, Fort Worth, Texas, United States

REFERENCES:
- [Result] Okeke CO, Quigley HA, Jampel HD, Ying GS, Plyler RJ, Jiang Y, Friedman DS. Adherence with topical glaucoma medication monitored electronically the Travatan Dosing Aid study. Ophthalmology. 2009 Feb;116(2):191-9. doi: 10.1016/j.ophtha.2008.09.004. Epub 2008 Dec 12. PMID 19084273